CLINICAL TRIAL: NCT05478421
Title: Https://Www.Zjuss.cn
Brief Title: Radiographic Bone Volume Alteration After Jaw Cyst Enucleation With Different Bone Grafts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Shi Jue, Doctor, The Dental Hospital of Zhejiang University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMSJC
Record Dates: First submitted 2022-06-21; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Jaw Cysts
MeSH Terms: conditions — Jaw Cysts

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Patients in control group will be treated by cyst enucleation.
- Collagen sponge group (Experimental): Cystic lesions in collagen sponge group will be filled by collagen sponge.
  Interventions: Procedure: Collagen sponge
- GBR group (Experimental): Cystic lesions in GBR group will be filled by deproteinized bovine substitute (DBBM, Bio-Oss®, granulometry 0.25-1 mm; Geistlich Pharma AG) and covered by absorbable collagen membrane (Bio-Gide®, Geistlich Pharma AG).
  Interventions: Procedure: GBR
- CS/GBR group (Experimental): Cystic lesions in GBR group will be filled by collagen sponge and deproteinized bovine substitute (DBBM, Bio-Oss®, granulometry 0.25-1 mm; Geistlich Pharma AG) and covered by absorbable collagen membrane (Bio-Gide®, Geistlich Pharma AG).
  Interventions: Procedure: CS/GBR

INTERVENTIONS:
Procedure: Collagen sponge — The bone cavity will be filled with collagen sponge.
  Arms: Collagen sponge group
Procedure: GBR — The bone cavity will be applied with guided bone regeneration with deproteinized bovine substitute (DBBM, Bio-Oss®, granulometry 0.25-1 mm; Geistlich Pharma AG) and absorbable collagen membrane (Bio-Gide®, Geistlich Pharma AG) .
  Arms: GBR group
Procedure: CS/GBR — The bone cavity will be applied with guided bone regeneration with collagen sponge and deproteinized bovine substitute (DBBM, Bio-Oss®, granulometry 0.25-1 mm; Geistlich Pharma AG) and absorbable collagen membrane (Bio-Gide®, Geistlich Pharma AG) .
  Arms: CS/GBR group

SUMMARY:
For decades, implantology has attracted extensive interest for restoration in patients with the defect of dentition. It has emerged as a very established prosthetic with a 5-year survival rate of 96% . However, defect of dentition resulted from jaw cyst remains an ongoing challenge for subsequent implantation treatment. Since it presents as a larger bone lesion than normal teeth extraction sockets and bone quality and quantity in teeth missing area can significantly impact dental implant failure rates .

Jaw cysts are one of the most common diseases occurring in the oral and maxillofacial area, and often cause destructive bone lesions followed by specific clinical features, such as located pain, swelling and loosen teeth. Over the years, enucleation of jaw bone cysts has been the standard method of management of jaw cysts because its conservational protocol to remove the lesion thoroughly and reserve important structures and functions. Unfortunately, management of the residual bony cavity remains as a huge dilemma whether to filing the defect with additional material. Clot formation in the first instance is the conventional option for residual cavity recovery. Iodoform sponges are traditionally used in cysts as stuffing material for inflammation preventative purpose, however, it cannot help with the following bone formation. Without any bone filling material, researches revealed that spontaneous bone healing index can be from 25.85% to 76% and from 43.46% to 81.03% after 6 and 12 months post-operative respectively. These ranged results indicated that spontaneous bone healing is not efficient enough especially for patients with the extraction of relevant teeth who may process a subsequent surgery for implantation. As an alternative to this, bone graft material in the surgery has gained increasing attention. Autogenous bone, artificial bone substitutes and mix of them are widely applied to achieve higher bone regeneration. Thereby an alternative surgical procedure should be considered for patients at risk of missing teeth because of jaw cysts. Whether bone graft material could make a remarkable improvement of bone regeneration after cyst enucleation and would this actually benefit the follow-up implantation? Answers are urged to be delivered.

Based on the published data, few studies have yielded in the bone healing comparison of spontaneous bone healing and xenograft in jaw cysts. Besides, with the development of medical radiograph, three-dimensional images have played a more important role in the clinic. Whereas, to our knowledge, most researches had adopted two-dimensional radiograph for measurement, such as panoramic radiographs rather than three dimensions.

Therefore, we conducted a prospective study to evaluate the shrinkage rate in cyst patients with different extra xenograft (Bio-Oss and collagen sponge). Cone beam computed tomography (CBCT) and three-dimensional model reconstruction were recommended for radiographic and digital analyzation. In summary, this study was aimed to evaluate bone volume augmentation after jaw cyst enucleation with different bone substitutes filling by CBCT and to analyze other influence factors for bone formation as well.

ELIGIBILITY:
Inclusion Criteria:

* jaw bone cyst with the maximum diameter from 1.5cm to 4.0cm;
* focal teeth were preserved with root canal treatment;
* no previous surgical treatment of the cyst site;
* no evidence of acute inflammation;
* in good physical status and oral health;
* regular attendance at control visits.

Exclusion Criteria:

* pregnancy or lactation;
* aggregate systemic pathologies such as diabetes, thyroid disorders, bone metabolism diseases, among others;
* patients taking calcium, bisphosphonates, glucocorticoids, or other drugs that can interfere with bone metabolism;
* patients with uncontrolled periodontal conditions, endodontic conditions and other oral disorders;
* heavy smoke (10 cigarettes/day or more).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Shrinkage rate of residual bone cavity | 3 months
  (pre-operative cyst volume - 3 / 6 months post-operative defect volume) / pre-operative cyst volume × 100%.
Shrinkage rate of residual bone cavity | 6 months
  (pre-operative cyst volume - 3 / 6 months post-operative defect volume) / pre-operative cyst volume × 100%.

SECONDARY OUTCOMES:
Bone density | 3 months
  HU value of newly-formed bone
Bone density | 6 months
  HU value of newly-formed bone

CONTACTS AND LOCATIONS:
Overall Officials: Jue Shi, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Berretta LM, Melo G, Mello FW, Lizio G, Rivero ERC. Effectiveness of marsupialisation and decompression on the reduction of cystic jaw lesions: a systematic review. Br J Oral Maxillofac Surg. 2021 Dec;59(10):E17-E42. doi: 10.1016/j.bjoms.2021.03.004. Epub 2021 Mar 23. PMID 34749963
- [Background] Buchbender M, Neukam FW, Lutz R, Schmitt CM. Treatment of enucleated odontogenic jaw cysts: a systematic review. Oral Surg Oral Med Oral Pathol Oral Radiol. 2018 May;125(5):399-406. doi: 10.1016/j.oooo.2017.12.010. Epub 2017 Dec 29. PMID 29396318
- [Background] Chiapasco M, Rossi A, Motta JJ, Crescentini M. Spontaneous bone regeneration after enucleation of large mandibular cysts: a radiographic computed analysis of 27 consecutive cases. J Oral Maxillofac Surg. 2000 Sep;58(9):942-8; discussion 949. doi: 10.1053/joms.2000.8732. PMID 10981973
- [Background] Chacko R, Kumar S, Paul A, Arvind. Spontaneous Bone Regeneration After Enucleation of Large Jaw Cysts: A Digital Radiographic Analysis of 44 Consecutive Cases. J Clin Diagn Res. 2015 Sep;9(9):ZC84-9. doi: 10.7860/JCDR/2015/13394.6524. Epub 2015 Sep 1. PMID 26501020